CLINICAL TRIAL: NCT02680249
Title: A Phase 1 Single Center, Open-Label, Randomized, Three-Way Crossover Study of the Relative Bioavailability of a Single Dose of CTP-656 in a Fasted, Fed Low-Fat and Fed Moderate-Fat Condition in Healthy Male Subjects
Brief Title: Food Effect Study of CTP-656 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CP656.1003
Record Dates: First submitted 2016-02-03; First posted 2016-02-11 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Safety, Bioavailability and Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CTP-656 Fed, low fat (Experimental): Single dose of CTP-656 150 mg administered after a low-fat breakfast
  Interventions: Drug: CTP-656
- CTP-656 Fasted (Experimental): Single dose of CTP-656 150 mg administered fasted
  Interventions: Drug: CTP-656
- CTP-656 Fed, high fat (Experimental): Single dose of CTP-656 150 mg administered after a moderate-fat breakfast
  Interventions: Drug: CTP-656

INTERVENTIONS:
Drug: CTP-656

SUMMARY:
Three way crossover study to assess the bioavailability of 656 under fed and fasted conditions.

DETAILED DESCRIPTION:
This study will assess in healthy male subjects a solid oral dose formulation of CTP-656 under fasted and fed conditions.

Primary:

• To characterize the relative bioavailability and pharmacokinetic profile of a single 150 mg solid oral dose of CTP-656 in healthy volunteers under fasted, fed low-fat and fed moderate-fat conditions.

Secondary:

* To characterize the pharmacokinetic profile of metabolites of CTP-656 following a single 150 mg solid oral dose of CTP-656 in healthy volunteers under fasted, fed low-fat and fed moderate-fat conditions.
* To assess the safety and tolerability following a single 150 mg solid oral dose of CTP-656 in healthy volunteers under fasted, fed low-fat and fed moderate-fat conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between 18 and 50 years of age, inclusive
* Body weight ≥ 50 kg and BMI within the range of 18 to 30 kg/m2, inclusive, at screening

Exclusion Criteria:

* History of clinically significant central nervous system (eg, seizures), cardiac, pulmonary, metabolic, renal (including nephrolithiasis), hepatic, including history of Gilbert's syndrome or gastrointestinal (GI) conditions
* PR interval ≥ 220 msec or QRS duration ≥ 120 msec or QTcF interval > 450 msec obtained at screening visit or prior to the first dose of study drug
* Liver function tests greater than the upper limit of normal.
* Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, or hepatitis C virus antibody at screening
* Urinalysis positive for greater than trace blood, protein or glucose
* A positive screen for alcohol, drugs of abuse, or tobacco use.
* Inability to comply with dietary restrictions during study participation.
* Donation or blood collection or acute loss of blood prior to screening.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Measurement of CTP-656 in plasma under fed and fasted conditions | 96 hours
  Geometric mean ratio of moderate-fat versus low-fat or fasted

CONTACTS AND LOCATIONS:
Overall Officials: Lana Pilja, Study Director — Concert Pharmaceuticals, Inc.
Locations (1):
- CMAX, Adelaide, South Australia, Australia